CLINICAL TRIAL: NCT00026182
Title: Randomized Phase II Study Of Interleukin-12 In Combination With Rituximab In Patients With Non-Hodgkin's Lymphoma
Brief Title: Rituximab and Interleukin-12 in Treating Patients With B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01865; NCI-2012-01865 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N0087; CDR0000068994; N0087 (Other: North Central Cancer Treatment Group); N0087 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Interleukin-12 Subunit p35; Interleukin-12

ARMS (2):
- Arm I (rituximab and recombinant interleukin-12) (Experimental): Patients receive rituximab IV on days 1, 8, 15, and 22. Patients receive interleukin-12 SC twice weekly beginning on day 2 and continuing until disease progression.
  Interventions: Biological: rituximab; Biological: recombinant interleukin-12; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment
- Arm II (rituximab and recombinant interleukin-12) (Experimental): Patients receive rituximab as in arm I. Patients are evaluated at week 12. Patients with stable or progressive disease receive interleukin-12 SC twice weekly until disease progression or for 24 weeks. Patients with a complete or partial response after rituximab are monitored until disease progression and then begin interleukin-12 SC twice weekly until further disease progression.
  Interventions: Biological: rituximab; Biological: recombinant interleukin-12; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Biological: recombinant interleukin-12 — Given SC
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Interleukin-12 may kill cancer cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Combining rituximab with interleukin-12 may kill more cancer cells. This randomized phase II trial is comparing how well giving rituximab together with two different schedules of interleukin-12 works in treating patients with B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the objective response in patients with B-cell non-Hodgkin's lymphoma treated with rituximab and 2 different schedules of interleukin-12*.

II. Compare the toxic effects of these regimens in these patients. III. Determine the objective response rate in patients with mantle cell lymphoma treated with these regimens.

IV. Determine the overall and progression-free survival of patients treated with these regimens.

V, Compare the quality of life of patients treated with these regimens. NOTE: *Interleukin-12 will no longer be available after 6/30/05.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to histology (mantle cell lymphoma vs other [closed to accrual as of 3/10/04]) and International Prognostic Factor Index (low and low-intermediate risk [closed to accrual as of 3/10/04] vs high-intermediate and high risk). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive rituximab IV on days 1, 8, 15, and 22. Patients receive interleukin-12* subcutaneously (SC) twice weekly beginning on day 2 and continuing until disease progression.

ARM II (closed to accrual as of 11/14/03): Patients receive rituximab as in arm I. Patients are evaluated at week 12. Patients with stable or progressive disease receive interleukin-12* SC twice weekly until disease progression or for 24 weeks. Patients with a complete or partial response after rituximab are monitored until disease progression and then begin interleukin-12 SC twice weekly until further disease progression.

NOTE: *Interleukin-12 will no longer be available after 06/30/05. Patients proceed to follow-up as outlined below.

Quality of life is assessed at baseline and at 3 and 6 months.

Patients are followed every 3 months for 1 year and then every 6 months for up to 4 years.

PROJECTED ACCRUAL: A total of 90 patients (45 per treatment arm [arm II closed to accrual as of 11/14/03]) will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20-positive B-cell non-Hodgkin's lymphoma
* Previously treated low-grade lymphoma considered incurable with standard therapy

  * Grade I or II follicular lymphoma*
  * Lymphoplasmacytic lymphoma*
  * Small lymphocytic lymphoma*
  * Nodal marginal zone lymphoma*
  * Extranodal marginal zone lymphoma of MALT type*
  * Splenic marginal zone lymphoma*
* Previously treated mantle cell lymphoma allowed
* Meets one of the following criteria for measurable disease:

  * Bidimensional diameter at least 1.5 cm by 1.5 cm on physical exam
  * At least 2 cm in one dimension by CT scan, MRI, or plain radiograph imaging
  * Palpable spleen at least 5 cm below the left costal margin
* No CNS involvement by lymphoma
* Performance status - ECOG 0-1
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* Creatinine ≤ 2 times ULN
* No New York Heart Association class III or IV heart disease
* No history of angina
* No uncontrolled peptic ulcer disease
* No uncontrolled infection
* No other active malignancy
* No autoimmune-related phenomena (e.g., antinuclear antibody less than 2 times ULN, rheumatoid factor less than 2 times ULN, and negative direct Coombs)
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Prior stem cell transplantation allowed
* More than 12 months since prior rituximab
* No prior interleukin-12
* No other concurrent immunotherapy
* Recovered from prior chemotherapy
* No concurrent chemotherapy
* No concurrent steroid therapy
* No concurrent radiotherapy
* Any number of prior therapies allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2001-10; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Objective response | 12 weeks
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. In addition, confidence intervals for the response probability will be calculated according to the approach of Duffy and Santner.
Objective response | 24 weeks
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. In addition, confidence intervals for the response probability will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Overall response rate for MCL patients | Up to 5 years
  Corresponding 95% confidence intervals will also be calculated.
Overall survival | From randomization to death due to any cause, assessed up to 5 years
  The distribution this time measure will be estimated using the method of Kaplan-Meier.
Time to treatment failure | From randomization to the treatment-specific definition of disease progression, death, or when the patient goes off study due to refusal or toxicity, assessed up to 5 years
  The distribution this time measure will be estimated using the method of Kaplan-Meier.
Complete response rate | Up to 5 years
  Will be assessed and descriptively summarized.
Quality of life assessed using FACT-BRM | Baseline
  Before and after treatment comparisons will be made using a paired samples t-test or its nonparametric equivalent. This two-sided test will have at least 80% power to detect a moderate effect size (0.42 times the standard deviation) in the FACT-BRM scores.
Quality of life assessed using FACT-BRM | 3 months
  Before and after treatment comparisons will be made using a paired samples t-test or its nonparametric equivalent. This two-sided test will have at least 80% power to detect a moderate effect size (0.42 times the standard deviation) in the FACT-BRM scores.
Quality of life assessed using FACT-BRM | 6 months
  Before and after treatment comparisons will be made using a paired samples t-test or its nonparametric equivalent. This two-sided test will have at least 80% power to detect a moderate effect size (0.42 times the standard deviation) in the FACT-BRM scores.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ansell, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States